CLINICAL TRIAL: NCT05764018
Title: Sex Differences in the Acute Effects of Caffeine Supplementation on Exercise in Normobaric Hypoxia
Brief Title: Caffeine and Hypoxia During Exercise in Males and Females
Acronym: HypoCaff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jozef Stefan Institute (Other)
Responsible Party: Principal Investigator, Tadej Debevec, Principal Investigator, Jozef Stefan Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HypoCaff
Record Dates: First submitted 2023-02-17; First posted 2023-03-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Caffeine; Hypoxia
Keywords: Caffeine; Hypoxia; Female physiology; Exercise
MeSH Terms: conditions — Hypoxia; Motor Activity | interventions — Caffeine; Sea Level Rise

STUDY DESIGN:
Intervention Model Description: Participants will perform four trials, to cover both levels of two factors; normoxia vs. hypoxia, and placebo vs. caffeine
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant will be blinded to both the supplement (placebo vs. caffeine) and the condition (normoxia vs. hypoxia). The investigator and the outcomes assessor will also be blinded to the supplement (placebo vs. caffeine), but both will be aware of condition (normoxia vs. hypoxia). Blinding success from the participants' perspectives will be assessed with an exit questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Normoxia-Placebo (Placebo Comparator): Participants will be breathing room air, and ingest a flavoured drink containing only a trivial amount of maltodextrin.
  Interventions: Other: Placebo; Other: Normoxia
- Normoxia-Caffeine (Experimental): Participants will be breathing room air, and ingest a flavoured drink containing a trivial amount of maltodextrin and 6 mg/kg body mass caffeine.
  Interventions: Dietary Supplement: Caffeine; Other: Normoxia
- Hypoxia-Placebo (Placebo Comparator): Participants will be breathing a 13% oxygen gas mixture, and ingest a flavoured drink containing only a trivial amount of maltodextrin.
  Interventions: Other: Hypoxia; Other: Placebo
- Hypoxia-Caffeine (Experimental): Participants will be breathing a 13% oxygen gas mixture, and ingest a flavoured drink containing a trivial amount of maltodextrin and 6 mg/kg body mass caffeine.
  Interventions: Dietary Supplement: Caffeine; Other: Hypoxia

INTERVENTIONS:
Dietary Supplement: Caffeine — Negligible amount of maltodextrin in flavoured drink solution containing 6 mg/kg body mass caffeine provided 45 minutes before exercise
  Arms: Hypoxia-Caffeine; Normoxia-Caffeine
Other: Hypoxia — Participants will be breathing from a hypoxic gas mixture (13% O2) for the duration of the exercise bout. This will simulate an altitude of approximately 3500 m.
  Other Names: Simulated altitude
  Arms: Hypoxia-Caffeine; Hypoxia-Placebo
Other: Placebo — Negligible amount of maltodextrin in flavoured drink solution provided 45 minutes before exercise.
  Other Names: No caffeine
  Arms: Hypoxia-Placebo; Normoxia-Placebo
Other: Normoxia — Participants will be breathing from ambient air (~21% O2) for the duration of the exercise bout. This will provide no hypoxic stimulus as the laboratory is located relatively near sea level (295 m)
  Other Names: Sea level
  Arms: Normoxia-Caffeine; Normoxia-Placebo

SUMMARY:
Several high-altitude destinations recommend their visitors to avoid caffeine, theoretically due to the associated diuresis which could contribute to acute mountain sickness. There is however no direct evidence for this association. In fact, caffeine ingestion is known to improve exercise performance at sea level, and may therefore help mountaineers during expeditions.

Sport science research is largely conducted in male participants, and the findings from these studies are assumed to apply to the female population. Given the known sex differences in body composition, hormones, and other physiological factors, this may not be appropriate. It is therefore important to conduct research in women, to allow for female-specific recommendations.

DETAILED DESCRIPTION:
As a result of transportation modernisation and tourism development, an increasing number of individuals are visiting high-altitude destinations for work and leisure purposes. The resulting exposure to (hypobaric) hypoxia is known to reduce exercise capacity due to a reduction in maximal oxygen uptake induced by lower oxygen pressure throughout the oxygen cascade. Several high-altitude destinations recommend their visitors to reduce or completely avoid caffeine intake during their stay. This recommendation is often based on the diuretic effects of caffeine, as the increased fluid loss through urine could accentuate dehydration, potentially contributing to feelings of acute mountain sickness. However, there is currently no scientific evidence to substantiate this recommendation. In fact, caffeine is known to be a particularly effective stimulant to improve exercise performance at sea level. Caffeine could therefore help mountaineers who engage in relatively intense physical activity during expeditions at altitude. The mechanisms underlying the ergogenic effects of caffeine are believed to originate centrally and peripherally. Of particular interest is the potential for caffeine to increase ventilation at submaximal and maximal exercise intensities. In a high-altitude environment, this could help to offset exercise- and hypoxia-induced hypoxemia, thereby enhancing exercise capacity.

Some studies have indeed provided evidence for the notion that caffeine could enhance exercise capabilities in hypoxia. Caffeine doses of 4.0 - 6.0 mg/kg body mass have been assessed, in (simulated and terrestrial) altitude environments equating to 2000 - 4300 m. In each case, it appeared that exercise performance and/or capacity at altitude could indeed be enhanced by caffeine ingestion. However, further mechanistic work is required, particularly in the assessment of the physiological effects of caffeine beyond typical exercise performance (time trial) and exercise capacity (peak power output, maximal oxygen uptake) outcomes. An enhanced holistic understanding of respiratory, cardiovascular, muscular and metabolic responses to exercise, caffeine and hypoxia is necessary to understand if caffeine ingestion at altitude is advisable.

Sport science research is largely conducted in male participants, and the findings from these studies are assumed to also apply to the female population. However, given the known sex differences in body composition, hormones, and other physiological factors, these assumptions may not be appropriate. It is therefore important to conduct research in women, to allow female-specific recommendations to be applied to athletes and to the general population.

As these are important considerations, the aim of this project is to investigate the effects of caffeine supplementation on exercise in hypoxia, and to determine whether these effects are influenced by sex differences.

24 healthy adult participants (12 male, 12 female) will be recruited to take part in the project. A preliminary testing session will be used to determine the maximal oxygen uptake of the participants in normoxia, and to familiarise them with the main trial protocol. A second preliminary laboratory visit will be used to measure the resting metabolic rate of the participants.

The main phase of the experiment will be a four-trial randomised crossover study; normoxia (ambient) vs. hypoxia (fraction of inspired oxygen = 0.13) and placebo (20 g maltodextrin) vs. caffeine (20 g maltodextrin + 6 mg/kg body mass caffeine). Participants will avoid caffeine, alcohol and intense exercise for 24 h prior to each laboratory visit. They will also replicate their diet for 24 h before each main trial. Each main trial will involve a 20-minute moderate-intensity cycling period, immediately followed by an incremental exercise test to exhaustion. Participants will be blinded to the environmental condition and the contents of the test drink. Outcome measures will include gas exchange variables, blood glucose/lactate concentration, muscle and brain oxygenation, blood oxygen saturation, heart rate and rating of perceived exertion. These measurements will provide a holistic overview of the broad physiological response to exercise, hypoxia and caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Regularly physically active (at least 30 mins of structured exercise 5 times per week).
* Sea-level natives.

Exclusion Criteria:

* presence of any medical risk factors to exercise and/or exposure to altitude
* presence of any medical condition that would make the protocol unreasonably hazardous for the participant
* smokers
* exposure to altitude above 2000 m in the last 2 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity. Self-identifying males and self-identifying females will be recruited for the study, and will form the two groups for comparison.
Enrollment: 29 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | Immediately prior to volitional exhaustion during the incremental exercise test
  Peak oxygen consumption (VO2peak, ml/kg/min) will be quantified from the end of each maximal exercise test and compared between groups and conditions.
Maximal aerobic power | At the instant of volitional exhaustion during the incremental exercise test
  Maximal aerobic power (MAP, W) will be quantified based on the time at which participants reach volitional exhaustion during the incremental exercise tests. This value will then be compared between groups and conditions.
Peak minute ventilation | Immediately prior to volitional exhaustion during the incremental exercise test
  Peak minute ventilation (VEpeak, L/min) will be quantified from the end of each maximal exercise test and compared between groups and conditions.
Peak heart rate | Immediately prior to volitional exhaustion during the incremental exercise test
  Peak heart rate (HRpeak, bpm) will be quantified from the end of each maximal exercise test and compared between groups and conditions.
Muscle oxygenation nadir | Immediately prior to volitional exhaustion during the incremental exercise test
  The nadir in muscle oxygenation (TSIMmin, %) will be quantified from the end of each maximal exercise test and compared between groups and conditions.
Peak blood lactate concentration | Immediately after volitional exhaustion during the incremental exercise test
  Blood lactate concentration will be measured immediately after the incremental exercise test to exhaustion ([BLapeak], mmol/L).

SECONDARY OUTCOMES:
Submaximal oxygen uptake | From the onset of exercise to the end of the submaximal exercise period at 20 minutes.
  Oxygen consumption (VO2, L/min) will be continuously monitored during the exercise bouts under each condition. Absolute oxygen uptake during the submaximal exercise phases will be compared between groups and conditions.
Submaximal minute ventilation | From the onset of exercise to the end of the submaximal exercise period at 20 minutes.
  Minute ventilation (VE, L/min) will be continuously monitored during the exercise bouts under each condition, and values during the submaximal exercise phases will be compared between groups and conditions.
Submaximal substrate oxidation | From the onset of exercise to the end of the submaximal exercise period at 20 minutes.
  Substrate oxidation, as respiratory exchange ratio (RER, arbitrary units) will be continuously monitored during the exercise bouts under each condition. The relative contributions of fat and carbohydrate will be estimated using this variable and compared between groups and conditions.
Submaximal muscle oxygenation | From the onset of exercise to the end of the submaximal exercise period at 20 minutes.
  Muscle oxygenation, as tissue saturation index (TSIM, %), will be continuously monitored during the exercise bouts under each condition using near-infrared spectroscopy. Absolute muscle oxygenation during the submaximal exercise phases, will be compared between groups and conditions.
Submaximal brain oxygenation | From the onset of exercise to the end of the submaximal exercise period at 20 minutes.
  Brain oxygenation, as tissue saturation index (TSIB, %), will be continuously monitored during the exercise bouts under each condition using near-infrared spectroscopy. Absolute brain oxygenation during the submaximal exercise phases, will be compared between groups and conditions.
Submaximal heart rate | From the onset of exercise to the end of the submaximal exercise period at 20 minutes.
  Heart rate (HR, bpm), will be continuously monitored during the exercise bouts under each condition. Absolute heart rate during the submaximal exercise phases, will be compared between groups and conditions.
Blood glucose concentration | At rest prior to exercise, and at the end of the submaximal exercise period at 20 minutes.
  Blood glucose concentration ([BG] mmol/L) will be measured at baseline and at the end of the submaximal exercise phase, to provide an indication of relative carbohydrate flux within each group and condition.
Blood lactate concentration | At rest prior to exercise, and at the end of the submaximal exercise period at 20 minutes.
  Blood lactate concentration ([BLa] mmol/L) will be measured at baseline and at the end of the submaximal exercise phase, to provide an indication of anaerobic metabolism within each group and condition.
Rating of perceived exertion | Every 5 minutes throughout the 20 minute submaximal exercise period.
  Ratings of perceived exertion will be measured throughout the submaximal exercise phases to establish the perception of workload, using a scale from 6 to 20 with higher values indicating a higher perception of exercise intensity. This will be compared between groups and conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Debevec, PhD, Principal Investigator — University of Ljubljana
Locations (1):
- University of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No